CLINICAL TRIAL: NCT00110877
Title: A Randomized, Controlled, Open-label Trial to Compare the Efficacy, Safety and Tolerability of TMC114/RTV Versus LPV/RTV in Treatment-Experienced HIV-1 Infected Patients
Brief Title: TMC114-C214: Trial of TMC114 Administered With Low Dose Ritonavir (RTV) in HIV-1 Infected Treatment Experienced Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002794; TMC114-C214 (Other: Tibotec Pharmaceuticals, Ireland); NCT00980902 (obsolete NCT alias)
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infection
Keywords: Human Immunodeficiency Virus; Treatment Experienced; TMC114-C214
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Experimental): LPV/rtv One 400mg LPV tablet twice daily with 100mg RTV
  Interventions: Drug: LPV/rtv
- 001 (Experimental): TMC114/rtv Two 300mg TMC114 tablets twice daily with 100mg RTV
  Interventions: Drug: TMC114/rtv

INTERVENTIONS:
Drug: LPV/rtv — One 400mg LPV tablet twice daily with 100mg RTV
  Arms: 002
Drug: TMC114/rtv — Two 300mg TMC114 tablets twice daily with 100mg RTV
  Arms: 001

SUMMARY:
Study TMC114-C214 is a randomized, controlled, open-label trial to compare the efficacy, safety and tolerability of TMC114 boosted with low dose ritonavir (RTV) versus Kaletra (LPV)/RTV in lopinavir-naïve treatment-experienced HIV-1 infected patients.

DETAILED DESCRIPTION:
Study TMC114-C214 is a randomized (patients are assigned to different treatment groups based on chance), controlled, open-label trial to compare the efficacy (effectiveness), safety and tolerability of TMC114 boosted with low dose ritonavir (RTV) versus Kaletra (LPV)/RTV in treatment-experienced HIV-1 infected patients. This research study will look at the safety of TMC114 and effectiveness in reducing the amount of HIV(viral load) in the blood. People included in this study will have received either Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) or Protease Inhibitors (PIs) or both. The duration of the study will be approximately 106 weeks, which includes a 4 to 6 week screening period, 96-week treatment period, and 4-week follow-up period. TMC114 300mg are orange tablets where 2 tablets are taken by mouth twice a day with 1 tablet of Ritonavir. Kaletra (LPV/RTV) is either a tablet or capsule taken twice a day. The oral capsule contains 133.3 mg LPV, 33.3 mg RTV and the film-coated tablet is available for oral administration in a strength of 200 mg of lopinavir and 50 mg of ritonavir. Dosing for all medication will occur for 96 weeks and you will be randomly assigned to either TMC114 or Kaletra.

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented HIV-1 infection
* Treatment with an Antiretroviral regimen (containing at least 2 NRTIs in combination with at least 1 NNRTI and/or 1 PI) for at least 12 weeks
* Plasma HIV-1 RNA >1000 copies/mL
* General medical condition does not interfere with the assessments and the completion of the trial

Exclusion Criteria:

* Patients for whom an investigational Antiretroviral is part of the current regimen, with the following exceptions if applicable (depending on local regulatory approval)
* tenofovir, emtricitabine, atazanavir, fosamprenavir
* Previous or current use of lopinavir, enfuvirtide (T-20), tipranavir and TMC114
* Life expectancy of less than 6 months
* Pregnant or breast-feeding
* Females of childbearing potential not willing to use effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 14 days after the end of the treatment period
* Patients with significantly decreased liver function or decompensation, irrespective of liver enzyme levels
* Participation in other investigational trials without prior approval of the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Viral load <400 copies/mL per TLOVR algorithm at Week 48 (Per Protocol Population) | 48 weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 96 weeks
Number of Participants With Viral load <400 copies/mL per TLOVR Algorithm at Week 96 (Per Protocol Population) | 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (103):
- United States (39):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Francisco, California
  - West Hollywood, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Orlando, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Berkley, Michigan
  - Camden, New Jersey
  - East Orange, New Jersey
  - Newark, New Jersey
  - The Bronx, New York
  - Durham, North Carolina
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Longview, Texas
  - Hampton, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Rosario
- Australia (4):
  - Darlinghurst
  - Melbourne
  - Perth
  - Surry Hills
- Vienna, Austria
- Belgium (2):
  - Antwerp
  - Brussels
- Brazil (6):
  - Curitiba
  - Distrito Barao Geraldo-Campina
  - Nova Iguaçu
  - Pinheiros
  - Rio de Janeiro
  - São Paulo
- Canada (4):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (2):
  - Providencia
  - Santiago
- Aalborg, Denmark
- France (4):
  - Nice
  - Paris
  - Rennes
  - Villejuif
- Germany (8):
  - Aachen
  - Berlin
  - Cologne
  - Düsseldorf
  - Hamburg
  - Mannheim
  - Osnabrück
  - Stuttgart
- Melissia-Athens, Greece
- Guatemala City, Guatemala
- Budapest, Hungary
- Malaysia (2):
  - Kuala Lumpur
  - Sungai Buloh
- Guadalajara, Mexico
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Rotterdam
- Panama City, Panama
- Portugal (2):
  - Lisbon
  - Porto
- San Juan, Puerto Rico
- Russia (5):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Volgograd
- South Africa (5):
  - Cape Town
  - Durban
  - Houghton, Johannesburg
  - Johannesburg
  - Pretoria
- Spain (2):
  - Barcelona
  - Madrid
- Zurich, Switzerland
- Thailand (2):
  - Bangkok
  - Khon Kaen
- London, United Kingdom

REFERENCES:
- [Result] Madruga JV, Berger D, McMurchie M, Suter F, Banhegyi D, Ruxrungtham K, Norris D, Lefebvre E, de Bethune MP, Tomaka F, De Pauw M, Vangeneugden T, Spinosa-Guzman S; TITAN study group. Efficacy and safety of darunavir-ritonavir compared with that of lopinavir-ritonavir at 48 weeks in treatment-experienced, HIV-infected patients in TITAN: a randomised controlled phase III trial. Lancet. 2007 Jul 7;370(9581):49-58. doi: 10.1016/S0140-6736(07)61049-6. PMID 17617272
- [Derived] Banhegyi D, Katlama C, da Cunha CA, Schneider S, Rachlis A, Workman C, De Meyer S, Vandevoorde A, Van De Casteele T, Tomaka F. Week 96 efficacy, virology and safety of darunavir/r versus lopinavir/r in treatment-experienced patients in TITAN. Curr HIV Res. 2012 Mar;10(2):171-81. doi: 10.2174/157016212799937218. PMID 22339125